CLINICAL TRIAL: NCT04724902
Title: The Effect of Elastic Bandage Compression on Pain and Function in Individuals With Knee Osteoarthritis - a Randomized Controlled Trial
Brief Title: The Effect of Elastic Bandage Compression on Pain and Function in Individuals With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Angélica Viana Ferrari, Principal Investigator (PT), Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE: 28484120.6.0000.5504
Record Dates: First submitted 2021-01-21; First posted 2021-01-26 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Knee Osteoarthritis
Keywords: Physiotherapy; Rehabilitation; Compression; Analgesia
MeSH Terms: conditions — Osteoarthritis, Knee; Agnosia | interventions — Compression Bandages

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial following guidelines from CONSORT (Consolidated Standards of Reporting Trials), TIDieR (Template for Intervention Description and Replication) and OARSI recommendations for clinical trials with patients with knee osteoarthritis.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The evaluations will be carried out by a "blind" evaluator with no information about the identification of the group to which the volunteer belongs.
  After the completion of the collections, the data will appear by a "blind" biostatistician, with no information on the identification of the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Compression Group (Experimental): The volunteer must remain supine on a stretcher, with both legs extended and relaxed. The intervention will be performed with elastic bandages (Selecta® of 13cm x 160 cm, composed of 45% cotton, 20% elastodiene and 27% polyamide) involving the entire knee surface, positioned considering anatomical aspects: covering the femoral condyles and the anterior tibial tuberosity). The bandage will involve the knee from the distal to the proximal, respecting the blood flow of the venous return. The level of compression was defined according to recommendations in the literature on compression interventions in lymphedema and venous changes, and should be kept between 30 mmHg and 60 mmHg. Variations on stipulated values may be interfered according to the volunteer's self-report, which should indicate a level of moderate, comfortable and pain-free compression. The intervention will be carried out for 20 minutes, once a day, for 4 consecutive days.
  Interventions: Other: Elastic bandage compression
- Sham Group (Sham Comparator): For Sham application, the volunteer must remain supine on a stretcher, with both lower limbs extended and relaxed. Elastic bandages will be used (Selecta® of 13cm x 160 cm, composed of 45% cotton, 20% elastodiene and 27% polyamide) involving the entire knee surface, positioned considering anatomical aspects: covering the femoral condyles and the anterior tibial tuberosity) . The bandage will involve the knee from the distal (tibial tuberosity) to the proximal (femoral condyles), respecting the blood flow of the venous return. However, in this group, no compression force will be performed, maintaining the pressure at 00 mmHg according to a previous reliability study. The procedure will be carried out for 20 minutes, once a day, for 4 consecutive days.
  Interventions: Other: Elastic bandage compression
- Control Group (No Intervention): The Control group will be composed of individuals with knee osteoarthritis, who make up the study's waiting list and will carry out evaluations at the same time intervals as the other groups, but will not receive any type of intervention and will be instructed not to start another treatment during their participation.

INTERVENTIONS:
Other: Elastic bandage compression — The compression will be applied with the volunteer in the supine position on a stretcher, with both lower limbs extended and relaxed. The intervention in the Compression group will be with elastic bandages involving the entire surface of the knee, positioned considering anatomical aspects: femoral condyles and the anterior tibial tuberosity. The level of compression must be maintained between 30 mmHg and 60 mmHg, according to the researched literature. The variations within these values will be stipulated according to the volunteer's self-report (comfortable and painless compression). The Shan Group will have the bandage wrapped around the knee without any compression force being exerted. The intervention will be carried out for 20 minutes, once a day, for 4 consecutive days. The Control group will be composed of volunteers who make up a study waiting list and will carry out the evaluations at the same time intervals as the other groups, but will not receive any type of intervention.
  Arms: Compression Group; Sham Group

SUMMARY:
Introduction and Purpose: Compression is a tactile stimulus that can reduce the perception of pain by stimulating tactile skin receptors and the speed of nerve conduction. It is highly associated with cryotherapy and other non-pharmacological physical agents without musculoskeletal pain control. However, there is still a lack of evidence on its possible effects on the modulation of this type of pain. This study will evaluate the effect of compression by elastic bandages, on pain and on the function of belonging with knee osteoarthritis (KO). Methodology: A randomized, blinded controlled clinical trial will be conducted. Individuals with KO (n = 90; both sexes; between 40 and 75 years old), will be allocated into three groups (n = 30 / group): Compression (submitted to compression by elastic bandage on the affected knee, 20 min, in 4 days consecutive); Sham (submitted to the same protocol with elastic bandage, but without compression); and Control (waiting list, without intervention). All will be taken one day before the start and one day after the last intervention. They will also be adopted in the 12th and 24th weeks after the intervention. The main outcome will be the pain intensity (Visual Analogue Scale). The Western Ontario & McMaster Universities Osteoarthritis (WOMAC) physical function questionnaire, physical function tests (step test, sit and stand test in 30s, 40m accelerated walk test), and the perception scale global change (GRC). Data analysis: SPSS 24.0 software will be used for descriptive analysis and performance of Kolmogorov-Smirnov tests, two-way ANOVA and multiple comparison tests. A 95% confidence level and a 5% significance level will be adopted.

DETAILED DESCRIPTION:
Study design: The study consists of a randomized controlled clinical trial that meets the guidelines recommended by CONSORT (Consolidated Standards of Reporting Trials) for non-pharmacological studies TIDieR (Template for Intervention Description and Replication) and OARSI recommendations for clinical trials with patients with knee osteoarthritis . The procedures will always be carried out at the same times for each volunteer, during the intervention and evaluation days, so that the same time interval between interventions and evaluations is respected.

The evaluations will be carried out by a "blind" evaluator with no information about the identification of the group to which the volunteer belongs. The evaluator will also be trained to maintain balance in discussions and questions raised by individuals regarding the research project and the interventions or evaluations used.

The screening, evaluation and intervention will be carried out at the School Health Unit - USE, Federal University of São Carlos (UFSCar), São Carlos. It is a non-probabilistic sampling study, for convenience and intentional. Volunteers will be recruited from public announcements and waiting lists from local and regional physiotherapy, rehabilitation, orthopedics and rheumatology outpatient clinics, as well as from an existing list of volunteers diagnosed with knee osteoarthritis, available in our laboratory.

Participants: 90 individuals will participate in the study, of both sexes, aged between 40 and 75 years, diagnosed with KO according to the clinical and radiographic criteria of the American College of Rheumatology. The individuals will perform a radiographic examination of both knees, with lateral, anteroposterior, and axial views. Radiographic exams will be performed at the University Hospital, UFSCar. The screening of volunteers will be carried out by a physiotherapist specialized in the subject and experienced in the evaluation of individuals with knee osteoarthritis.

Ethical aspects: The project was initially submitted to the Ethics and Research Committee involving human beings (Plataforma Brasil), approved under Opinion Number: 3.955.692, and submitted to the registration of clinical trials (www.clinicaltrials.gov). Then, the study activities will be carried out. Volunteers will receive a verbal and written explanation of the objectives and methodology of the study, and those who agree to participate will sign an informed consent form.

Randomization: The individuals included in the study will be stratified by sex and randomly divided using the digital tool (www.randomization.com). Three groups will be randomized, with 30 individuals each: a) Compression: compression will be applied around the entire knee with KO through tensioned elastic bandages; b) Sham will also receive the application of elastic bandages around the knee with KO, but without compression; c) Control: patients on the waiting list, who will not receive intervention. To avoid selection bias, the confidential allocation method will be adopted using an opaque, non-translucent and sealed envelope. In addition, the group to which the individual belongs will only be revealed immediately before the intervention.

Sample size: The sample size was calculated preliminarily using the G * Power software (version 3.1.3; University of Trier, Germany). Two calculations were performed, the first considering pain (assessed by VAS) and the second, function (assessed by the WOMAC questionnaire). The calculation was based on the application of an F-test for the difference between three independent means (three groups). The effect size considered for this calculation, based on a previous study, was d = 0.45 for VAS, and d = 0.39 for WOMAC, which after conversion represent respectively f = 0.225 and f = 0.195). The effect sizes of f are between small and moderate, and match the rating range for the displayed d values. The level of significance was 5% and the power 95%. The calculations indicated a total of 54 individuals by the VAS and 72 individuals by the WOMAC questionnaire. The calculation to be considered will be related to the WOMAC questionnaire, with 24 individuals per group, making a total of 72 individuals. Considering a possible dropout rate of 20%, 29 participants must be allocated to each group, but to facilitate calculations and randomization, 30 participants will be allocated per group, totalling 90 individuals included in the study. A more reliable calculation will be performed after a preliminary analysis of the data collected from a pilot study.

Intervention: The elastic bandages used will be (Selecta® 13cm x160 cm, composed of 45% cotton, 20% elastodiene and 27% polyamide) involving the entire knee surface, positioned considering anatomical aspects: covering the femoral condyles and the anterior tuberosity of the tibia. The bandage will involve the knee from the distal (tibial tuberosity) to the proximal (femoral condyles), respecting the blood flow of the venous return. The level of compression was defined according to recommendations in the literature on compression interventions in lymphedema and venous changes, and should be kept between 30 mmHg and 60 mmHg. The occurrence of any sign of venous stasis (flushing and / or edema) may also indicate the need for a reduction in the level of compression or interruption of the procedure.

To standardize the level of compression presented, a previous reliability study (n = 10) was performed, with the aid of a pressure gauge (Stabilizer® - Chattanooga Group), positioned on the knee, between the patient's skin and the elastic bandage . The manometer was inflated to 40mmHg, a value indicated by the manufacturer as the resting pressure of the pneumatic bag47, and we then began to wrap the knee with the bandage. The number of turns that the tensioned elastic bandage allowed to wrap the knee was collected to reach the indicated compression range (30 mmHg ≤ x ≥ 60 mmHg), and if necessary, more than one band could be used. It was also evaluated what level of compression the Sham group would receive with the non-tensioned bandage. In both groups, the circumference of the knees was collected at three points (popliteal fossa, 10 cm above and 10 cm below) and the number of turns that were taken with the bandage.

This first step was performed in the test-retest format, with an interval of seven days, so that it was possible to calculate the intra-rater reliability level, which indicated a Kappa Coefficient48 of 0.625, considered a substantive agreement. From the reliability study, it was possible to calculate the average number of turns that should be performed both in the Compression group and in the Sham group so that the level of compression is maintained in the stipulated range. In the Compression group, all patients used a bandage, with an average of 5.7 turns (ranging from 5 to 7 turns) and the pressure level maintained at 48 mmHg (ranging from 46 to 52 mmHg). In the Sham group, everyone also used a bandage, with an average of 4 turns (ranging from 3 to 5 turns) and the pressure level maintained at 00 mmHg.

After the completion of the evaluations, the individuals of the three groups will receive face-to-face training, consisting of therapeutic exercises recommended for the treatment of knee osteoarthritis (KO), as well as a booklet with the proposed exercises, prepared by our research group, so that they can also perform the exercises without supervision. After completing the evaluations, participants in the Sham and Control groups will be able to receive the same treatment available to the Compression group, if they so request. In addition, they will remain on our list of volunteers for further studies in KO. The applications of the interventions will be performed by a physiotherapist previously trained on these procedures performed on the knee joint. The therapist will also be trained to maintain balance in explaining the study's general outlook, in discussions and questions raised by individuals about the research project and about the interventions or assessments used.

Data analysis: The registration of the data collected in the evaluations will be carried out through digital forms (Google Forms) and automatically stored in an electronic database in the Cloud (Google Drive), protected by password, to guarantee the security of the data and the participants. After completion of the collections, the data will be analysed by a "blind" biostatistician, with no information on the identification of the groups, using the SPSS 24.0 software (SPSS Inc, Chicago, IL).

The independent variables of interest in the study are group (Compression, Sham and Control) and time [pre- (assessment 1) and post-intervention (assessments 2, 3 and 4)]. The dependent variables are VAS (pain intensity), WOMAC (total score), Step test (seconds), Sit and stand test in 30 seconds (number of repetitions), and 40 m accelerated walk test (speed in m / s). The data distribution, or normality, will be tested by the Kolmogorov-Smirnov test and, according to the result, parametric or non-parametric tests will be used.

Initially, descriptive analyses will be performed, using measures of central tendency and dispersion: mean and standard deviation when following a normal distribution, and the median, minimum and maximum, when non-normal distribution. For normal data, the two-way ANOVA with mixed design will be the parametric test chosen to compare the means of the dependent variables, considering both factors simultaneously, one from repeated measurements (pre- and post-intervention, and follow up of 12 and 24 weeks) and another of independent samples (Compression, Sham and Control). If significant differences are found, tests of multiple comparisons (Post-Hoc) will be performed to assess the differences. For distribution of non-normal data, the possible reasons for non-normality, analysis of possible correction and then non-parametric tests can be applied, using both repeated (time) and non-repeated (groups) comparisons with Bonferroni adjustments or similar.

For all variables, a 95% confidence level will be determined and a significance level of 5% will be considered statistically significant. Added to this, the difference between the groups will be compared to the MDCI values defined for each variable. When the MDCI values are not available, Cohen's d coefficient will be calculated (effect size:> 0.8 large, close to 0.5 moderate and ≤ 0.2 small). Finally, to preserve the benefit of randomization, allowing for a balanced distribution of prognostic factors in the compared groups and, consequently, the observed effect, an intention-to-treat analysis will be adopted using the expectation-maximization imputation method.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of knee osteoarthritis according to the clinical and radiographic criteria of the American College of Rheumatology: signs of osteoarthritis in at least one of the compartments of the knee joint (tibiofemoral and / or in the patellofemoral joint); grade 2 or 3, according to Kellgren & Lawrence criteria in the radiographic examination;
* Minimum score of 04 cm on the Visual Analogue Scale (EVA, total of 10 cm);
* Accept and sign the informed consent form.

Exclusion Criteria:

* Regular practice of moderate or intense physical activity for more than 45 minutes a week;
* Having started physical activity or undergone any physical therapy treatment in the previous 3 months;
* Use of corticosteroid infiltration in the knee (previous 6 months);
* Performing previous surgery on the knee or hip;
* Presence of some clinical restriction that makes it impossible for them to participate in the proposed evaluations or interventions (cardiorespiratory, neurological, musculoskeletal, vascular changes, and / or the presence of skin lesions when applying the bandage).

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline - Visual Analog Scale (VAS) | Baseline, immediately after intervention and follow-up evaluations of 12 and 24 weeks.
  The scale will be made available visually to the individual so that he can classify the intensity of the average pain relative to the last week, and also before and after the performance of each functional physical test. The scale will vary from 0 to 10 cm, with 0 being the complete absence of pain, and 10 being the maximum pain intensity reported by the individual. The 1.75cm reduction will be considered an MDCI.
Change from baseline WOMAC (Western Ontario e o McMaster Universities Osteoarthritis Index) - Pain scale | Baseline, immediately after intervention and follow-up evaluations of 12 and 24 weeks.
  Self-report questionnaire, designed to assess problems experienced by individuals with lower limb OA, in the last 72 hours. The volunteer will be asked to answer 24 questions, which comprise three domains: pain, stiffness and physical function. The scores for the items are expressed using the Likert scale, classified as: none = 0, low = 25, moderate = 50, severe = 75 and very severe = 100. Higher scores indicate higher levels of pain, stiffness and physical dysfunction . The reduction of 8.74 points in the pain domain, from the baseline, will be considered an MDCI.

SECONDARY OUTCOMES:
Change from baseline WOMAC (Western Ontario e o McMaster Universities Osteoarthritis Index) - stiffness and physical dysfunction scales | Baseline, immediately after intervention and follow-up evaluations of 12 and 24 weeks.
  Self-report questionnaire, designed to assess problems experienced by individuals with lower limb OA, in the last 72 hours. The volunteer will be asked to answer 24 questions, which comprise three domains: pain, stiffness and physical function. The scores for the items are expressed using the Likert scale, classified as: none = 0, low = 25, moderate = 50, severe = 75 and very severe = 100. Higher scores indicate higher levels of pain, stiffness and physical dysfunction . The 12% improvement over the initial assessment will be considered a MDCI.
Sit and stand test - 30 seconds | Baseline, immediately after intervention and follow-up evaluations of 12 and 24 weeks.
  The test will be performed using an armless chair, with a seat height of approximately 43 cm from the floor. The chair will be positioned with the back against a wall to prevent oscillations and will have non-slip rubbers under its supports. The participant will sit in the chair, with the back straight, feet apart, aligned with the width of the shoulders and supported on the floor at an angle slightly behind the knee line. The arms should remain crossed against the chest and to aid in balance, one foot may remain slightly in front of the other.
  The test will last 30 seconds and in that time the number of complete cycles that the individual performs will be counted, that is, how many times he moves from sitting to standing and sits down again. Scores can range from 0, for those who cannot complete a single cycle, to values greater than 20 repetitions, for the most physically fit individuals. The increase of 2 complete cycles will be considered an MCDI.
Step test | Baseline, immediately after intervention and follow up evaluations of 12 and 24 weeks.
  The test will consist of going up and down, uninterruptedly, a flight of stairs with 9 steps, located in a bright and wide environment. Each step will be 20 cm high and it will be allowed to use the handrail as a safety tool. The individual will be positioned in front of the stairs, and by voice of command he will be guided to go up the 9 steps and descend right afterwards, returning to the starting point.
  departure, and thus will end the test. The score will be calculated by counting the time, in seconds, that the volunteer fulfills the test. A minimum detectable difference (MDD) will be considered for a reduction of 5.5 seconds in the test execution.
40 meter accelerated walk test (4x10m) | Baseline, immediately after intervention and follow up evaluations of 12 and 24 weeks.
  Participants will be asked to walk as fast, safely, without running, a distance of 10 m from a cone, then perform a half turn in a second cone, return and repeat the process up to the 40 meter mark covered . The test score will be based on the gait speed performed by the individual, and the higher the speed, the better the result. The speed will be obtained through the distance traveled data (40 meters) and the time, in seconds, needed to complete the route. The increase of 0.2 m / s will be considered an MCDI.
Global rating of change - GRC scale | Immediately after intervention and follow up of 12 and 24 weeks.
  Its use has been recommended for the outcome of chronic pain, mainly in clinical trials aiming at better applicability of the results in clinical practice. It is used to quantify the patient's improvement or worsening over time, according to the patient's perception. The volunteer will be asked to assess their health status. current, associated with knee pain, compared to the pre-intervention period. It consists of a numerical analog scale, which quantifies the patient's self-perception of improvement after the application of an intervention. The scale has a total of 15 points, and ranges from -7 (much worse) to +7 (much better). For this variable, an increase of 2 points will be considered an MCDI. In addition, studies have indicated that, considering the Minimum Important Difference (MID), variations of 1 to 3 points may indicate small changes, 4 or 5 as moderate changes and 6 or 7 as large changes.

OTHER OUTCOMES:
Blinding and use of elastic bandage. | Follow up 24 weeks
  In the last evaluation, participants in the sham and compression groups will be asked if they believe they have received the treatment, so that the effectiveness of the blinding strategy could be verified. In addition, it was questioned whether these volunteers continued to use the elastic bandage and how often they did so.

CONTACTS AND LOCATIONS:
Locations (1):
- Angelica Viana Ferrari, São Carlos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The registration of the data collected in the evaluations will be carried out by means of digital forms and automatically stored in an electronic database in the Cloud, protected by password, to guarantee the security of the data and the participants. The project manager and the research assistant will regularly monitor the study data sets and make recommendations on how necessary protocol modifications or the termination of all or part of the study. The data of the participants that substantiate the results reported in this article will be shared after masking (text, tables, figures, appendices), immediately after publication. In addition, the study protocol and the clinical trial report (both with the planned statistical analysis) will be made available by the researchers who proposed the methodology. Data requests or any form of analysis should be sent to ferrari.angelicaviana@gmail.com or tania@ufscar.br. Requesters must sign a data access agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Participant data that underlie the results reported in this paper will be shared after blinding (text, tables, figures, appendices), immediately following publication.
Access Criteria: Request for data or any form of analysis should be directed to ferrari.angelicaviana@gmail.com or tania@ufscar.br. Requesters will be asked to sign a data access agreement.

REFERENCES:
- [Derived] Ferrari AV, Perea JPM, Dantas LO, Silva HJA, Serrao PRMDS, Sendin FA, Salvini TF. Effect of compression by elastic bandages on pain and function in individuals with knee osteoarthritis: protocol of a randomised controlled clinical trial. BMJ Open. 2022 Nov 16;12(11):e066542. doi: 10.1136/bmjopen-2022-066542. PMID 36385041